CLINICAL TRIAL: NCT04393922
Title: Spasticity After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Monica Perez, Scientific Chair Arms + Hands Lab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00212201
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury, Spasticity, TMS
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 (Experimental): To accomplish this aim, we will conduct one experiment in two sessions separated by 2- 3 days using a crossover design. Participants will be assigned into one of three groups: spastic SCI, non-spastic SCI, and controls. We expect that people enrolled in Aim 1 will complete 2 visits within 1 week.
  Visit 1 Measurements:
  * MVCs
  * MEP Recruitment Curves
  * iMEPs
  * StartReact
  Visit 2 Measurements:
  * Participant Reported Spasticity
  * MAS
  * PSAD
  * KINARM
  * MRI of brain and spinal cord
  Interventions: Behavioral: Acoustic stimuli (Startle)
- Aim 2 (Experimental): To accomplish this aim, we will use a randomized crossover design study with spastic SCI participants receiving a single intervention combining non-invasive acoustic stimuli (Startle) or sham-Startle with motor training to enhance cortico- and reticulo-spinal contribution, separated by ~2 weeks.
  Visit 1 and Visit 2
  Single intervention of:
  Startle + exercise training OR sham-Startle + exercise training
  Pre and post measurements:
  * MVCs
  * MEP recruitment curves
  * iMEPs
  * StartReact
  * Participant reported spasticity
  * MAS
  * PSAD
  * KINARM
  * Neuromechanical hand and/or leg testing
  * GRASSP
  * TRI-HFT
  * 10-meter walk test
  * Pendulum Test
  Interventions: Behavioral: Acoustic stimuli (Startle)

INTERVENTIONS:
Behavioral: Acoustic stimuli (Startle) — A startle stimulus (120 dB, 500 Hz, 50 ms) will be delivered through headphones

SUMMARY:
Very often, people who have a SCI have difficulty doing things with their arms or hands as a result of muscle stiffness , or spasticity. Spastacity can cause problems performing even the simplest of everyday tasks. This research will help us understand how the body recovers and changes neurologically after SCI.

DETAILED DESCRIPTION:
After spinal cord injury (SCI), damage to descending motor pathways has been associated with the development of spasticity (Frigon and Rossignol, 2006; Trompetto et al., 2014). Self-reported questionnaires and clinical exams indicate that individuals with incomplete SCI, who showed residual descending connectivity, have a high prevalence of spasticity compared to individuals with complete SCI (Little et al., 1989; Holtz et al., 2017). In agreement, our recent electrophysiological and spinal cord imaging data in humans with a diagnosis of a clinically motor complete SCI showed the presence of descending motor pathway connectivity in individuals with spasticity compared to those without spasticity (Sangari et al., 2019). However, which descending motor pathways influence spasticity following SCI, and to what extent, remains poorly understood. This proposal has two main goals: 1) to examine the contribution of cortico- and reticulo-spinal pathways to spasticity in upper and lower limb muscles, and 2) to develop strategies to promote functional recovery of upper and lower limb spastic muscles in humans with chronic incomplete SCI. The aims below will test two main hypotheses.

In Aim 1, we will use transcranial magnetic stimulation and startle acoustic stimuli to examine the contribution of the cortico- and reticulo-spinal pathway to upper and/or lower limb muscles electromyographic activity. Spinal cord atrophy and morphological characterization of cortico- and reticulo-spinal pathways will be assessed with high-resolution magnetic resonance imaging. Physiological and neuroimaging outcomes will be associated with clinical assessment of spasticity.

In Aim 2, we propose to enhance cortico- and reticulo-spinal contribution to upper and/or lower limb function in spastic muscles by using a novel intervention combining startle acoustic stimuli with motor training.

This research will provide new knowledge about the contribution of descending motor pathways to the control of spasticity in upper and lower limb muscles following incomplete cervical SCI (Aim1) and might lead to the development of a novel rehabilitation intervention to improve upper and lower limb motor function recovery by enhancing residual descending control over spinal networks (Aim 2).

ELIGIBILITY:
Inclusion criteria for individuals with SCI

* Chronic SCI (≥1 year of injury)
* Incomplete spinal cord injury at T12 or above
* Males and Females
* Ages 18-75 years

Inclusion criteria for non-spastic individuals with SCI

-MAS scores of 0 and 1

Inclusion criteria for spastic individuals with SCI

* MAS scores of 2, 3 and 4
* The ability to perform a voluntary flexion and extension of the elbow and/or knee or ankle
* The ability to reach and grasp an object

Inclusion criteria for health controls

* Males and females
* Ages 18-75 years
* Right-handed
* Able to perform elbow and/or knee or ankle flexion and extension

Exclusion Criteria for individuals with SCI and healthy controls:

* Uncontrolled medical problems including pulmonary, cardiovascular, or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Pacemaker
* Metal plate in skull
* History of seizures
* Receiving drugs acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
* Pregnant females
* Ongoing cord compression or a syrinx in the spinal cord or who suffer from a spinal cord disease such as spinal stenosis, spina bifida, or herniated cervical disk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-06-18 (Estimated); Study Completion 2024-05-18 (Estimated)

PRIMARY OUTCOMES:
MEP recruitment curves | 3-4 hours
  Ten stimuli (0.2 Hz) will be delivered at each intensity to plot the mean peak-to-peak amplitude of the MEP from the non-rectified response against the TMS intensity in each subject (MEP recruitment curve).
Ipsilateral MEPs (iMEPs) | 3-4 hours
  Ten stimuli will be delivered during head straight and ten stimuli will be delivered during lateral head rotation, randomly alternated (0.2 Hz).
StartReact | 3-4 hours
  Here, participants will be asked to observe a light-emitting diode (LED) located in front of their head. When the LED will illuminate, individuals will be asked to move their arm or leg. In some trials, the LED will be presented with either a quiet acoustic stimulus (80 dB, 500 Hz, 50 ms) or a startling acoustic stimulus (SAS, 120 dB, 500 Hz, 50 ms) delivered through a headphone.
Participant reported spasticity | 3-4 hours
  Spasticity questionnaire
Modified Ashworth Scale (MAS) | 3-4 hours
  This scale measures resistance encountered during manual passive muscle stretching using a six-point ordinal scale.
Portable Spasticity Assessment Device (PSAD)' | 3-4 hours
  The PSAD combine biomechanical and electrophysiological measurements for an objective quantification of active and passive component of muscle stiffness
Pendulum Test | 3-4 hours
  As part of the physical exam, we will use the pendulum test to measure muscle tone at the knee by using gravity to provoke muscle stretch reflexes during passive swinging of the lower limb.
10-meter walk test | 3-4 hours
  10-meter walk test will be used to assess walking speed
Graded and Redefined Assessment of Strength, Sensibility and Prehension (GRASSP). | 3-4 hours
  This exam measures clinical impairment that incorporates three domains vital to upper-limb function: sensation, strength, and prehension.
Toronto Rehabilitation Institute-Hand Function Test (TRI-HFT) | 3-4 hours
  This exam measures gross motor function frequently used to manipulate objects that participants may encounter in their daily lives.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No